CLINICAL TRIAL: NCT04223466
Title: Video-assisted Thoracoscopic Thymectomy Versus Subxiphoid Thymectomy: Short- Term and Long- Term Results
Brief Title: Video-assisted Thoracoscopic Thymectomy Versus Subxiphoid Procedure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Subxiphoid ZYP1
Record Dates: First submitted 2020-01-08; First posted 2020-01-10 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Thymectomy
Keywords: Video-assisted thoracoscopic surgery; Subxiphoid approach

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subxiphoid group (Experimental): Subxiphoid procedure for thymectomy.
  Interventions: Procedure: Subxiphoid surgery procedure
- VATS group (Active Comparator): Video-assisted thoracoscopic thymectomy through chest wall.
  Interventions: Procedure: VATS surgery procedure

INTERVENTIONS:
Procedure: Subxiphoid surgery procedure — Subxiphoid procedure for thymectomy
  Arms: Subxiphoid group
Procedure: VATS surgery procedure — VATS procedure for thymectomy
  Arms: VATS group

SUMMARY:
Surgerys used in thymectomy for myasthenia gravis and anterior mediastinal tumours have become much less invasive in recent years. In our study, the surgical technique which resected the thymus below the xiphoid process and the technique which was regarded as conventional video- assisted thoracoscopic surgery (VATS) thymectomy was compared.

ELIGIBILITY:
Inclusion Criteria:

1. Thymoma with or without myasthenia gravis；
2. Generalized myasthenia gravis not sensitive to conservative medicine treatment;
3. Good cardiopulmonary function.

Exclusion Criteria:

1. Cardiopulmonary function can't bear surgery;
2. Generalized myasthenia gravis with MuSK(+).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale of postoperative pain | within 3 days
  in score
Operation time | one day
  in minutes
The amount of blood loss | one day
  in milliliter
Duration of drainage | with 7 days
  in days
Duration of hospital stay | with 7 days
  in days

SECONDARY OUTCOMES:
Complete remission rates | 5 years
  Complete remission rates after 5 year follow-up of thymectomy for myasthenia gravis
Recurrence rate | 5 years
  Recurrence rate after 5 year follow-up of thymectomy for thymoma
Overall survival | within 10 years
  Overall survival in rate

CONTACTS AND LOCATIONS:
Locations (1):
- Yunpeng, Jinan, Shandong, China